CLINICAL TRIAL: NCT06610071
Title: Near-infrared Fluorescence Image-guided Surgery for Malignant Soft Tissue Tumor With Low-dose Second Window Indocyanine Green Technique: a Multicenter Randomized Controlled Trial
Brief Title: NIFR Image-guided Surgery for Malignant Soft Tissue Tumor With Low-dose SWIG Technique
Acronym: NIFR;SWIG
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Plastic Surgery Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College (Other)
Collaborators: 1、 Department of Plastic and Reconstructive Surgery, Peking University Third Hospital (Unknown); 2、 Department of Plastic and Reconstructive Surgery, 1st Medical Center of Chinese PLA General Hospital (Unknown); 3、 Department of Plastic and Reconstructive Surgery, Peking University International Hospital (Unknown)
Responsible Party: Principal Investigator, Lei Cui, Principal Investigator, The Plastic Surgery Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CFH2024-2-4043
Record Dates: First submitted 2024-09-01; First posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Dermatofibrosarcoma Protuberans (DFSP); Skin Squamous Cell Carcinoma
Keywords: near-infrared fluorescence imaging; second window indocyanine green; dermatofibrosarcoma protuberans; skin squamous cell carcinoma
MeSH Terms: conditions — Dermatofibrosarcoma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Patients with DFSP in the first experimental group (Experimental): The ICG was injected intravenously 24 hours before surgery at a dose of 0.25 mg/kg in the first experimental group.
  Interventions: Drug: ICG administration
- Patients with DFSP in the second experimental group (Experimental): The ICG was injected intravenously 24 hours before surgery at a dose of 25 mg/patient in the second experimental group.
  Interventions: Drug: ICG administration
- Patients with DFSP in the control group (No Intervention)
- Patients with sSCC in the first experimental group (Experimental): The ICG was injected intravenously 24 hours before surgery at a dose of 0.25 mg/kg in the first experimental group.
  Interventions: Drug: ICG administration
- Patients with sSCC in the second experimental group (Experimental): The ICG was injected intravenously 24 hours before surgery at a dose of 25 mg/patient in the second experimental group.
  Interventions: Drug: ICG administration
- Patients with sSCC in the control group (No Intervention)

INTERVENTIONS:
Drug: ICG administration — The ICG was injected intravenously 24 hours before surgery at a dose of 0.25 mg/kg in the first experimental group.
  Arms: Patients with DFSP in the first experimental group
Drug: ICG administration — The ICG was injected intravenously 24 hours before surgery at a dose of 25 mg/patient in the second experimental group.
  Arms: Patients with DFSP in the second experimental group
Drug: ICG administration — The ICG was injected intravenously 24 hours before surgery at a dose of 0.25 mg/kg in the first experimental group
  Arms: Patients with sSCC in the first experimental group
Drug: ICG administration — The ICG was injected intravenously 24 hours before surgery at a dose of 25 mg/patient in the second experimental group.
  Arms: Patients with sSCC in the second experimental group

SUMMARY:
This research study will evaluate how near-infrared fluorescence (NIRF) imaging with low-dose second window indocyanine green (ICG) can assist in the radical resection and pathologic diagnosis of malignant soft tissue sarcoma, such as dermatofibrosarcoma protuberans (DFSP) and skin squamous cell carcinoma (sSCC) during surgery.

DETAILED DESCRIPTION:
To improve the accuracy of radical resection by reducing the risk of missed diagnosis of positive margin, this study will explore clinical application of near-infrared fluorescence imaging with modified low-dose SWIG technique in guiding radical resection of malignant soft tissue tumor. The investigators conduct a multi-center, multi-subgroup, prospective randomized controlled trial. The participants will be first stratified according to histological type involving dermatofibrosarcoma protuberans (DFSP) and skin squamous cell carcinoma (sSCC). The patients with DFSP or sSCC will be then randomly assigned to three groups. Patients in the control group will not receive ICG administration. The ICG was injected intravenously 24 hours before surgery, at a dose of 0.25 mg/kg in the first experimental group and 25 mg/patient in the second experimental group, respectively. The patients in the control groups will undergo traditional assessment of surgical margins.The patients in the experimental groups, on the other hand, will be scheduled to intraoperative near-infrared fluorescence imaging to scan gross tumor, tumor bed and cross-sectional specimen. The 2-year local recurrence rate will be regarded as primary outcome. The number of positive margins will be compared among groups. The investigators will also calculate the sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV) with 95% confidence intervals based on fluorescent signal of tumor bed in the experimental groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients with DFSPs or sSCC in heads, extremities or trunk

Exclusion Criteria:

* seafood/iodine allergy
* hyperthyroidism
* pregnancy
* myasthenia gravis
* acute severe hypertension

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 592 (Estimated)
Dates: Start 2024-10-30 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
2-year local recurrence rate | up to 24 months

SECONDARY OUTCOMES:
number of positive margins | through study completion, an average of 2 years
sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV) | through study completion, an average of 2 years
Adverse effects | through study completion, an average of 2 years

IPD SHARING:
Plan to Share IPD: Yes
The IPD will include patient characteristics, tumor location, tumor size and histological type and grade. The number of positive margins will be recorded. The sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV) will also be calculated. The adverse effects between first and second experimental groups will be compared. The 2-year local recurrence rate will be viewed as primary outcome.
Supporting Information: Study Protocol

REFERENCES:
- See also: Related Info — https://www.frontiersin.org/journals/surgery/articles/10.3389/fsurg.2022.984857/full